CLINICAL TRIAL: NCT02269930
Title: An Open-label Crossover Phase 1 Study to Evaluate the Pharmacokinetic Profiles of BIIB017 (Peginterferon Beta-1a) and Rebif® (Interferon Beta-1a) in Healthy Volunteers
Brief Title: Study to Evaluate the Pharmacokinetic Profiles of BIIB017 (Peginterferon Beta-1a) and Rebif® (Interferon Beta-1a) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 105HV105
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — peginterferon beta-1a; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Treatment Sequence 1: Single subcutaneous (SC) dose of BIIB017 on Day 1; and SC doses of Rebif on Days 29, 32, 34, 36, 39, and 41 Treatment Sequence 2: SC doses of Rebif on Days 1, 4, 6, 8, 11, and 13; and a single SC dose of BIIB017 on Day 29
  Interventions: Drug: peginterferon beta-1a; Drug: Rebif
- Group 2 (Experimental): Treatment Sequence 1: SC doses of Rebif on Days 1, 4, 6, 8, 11, and 13; and a single SC dose of BIIB017 on Day 29 Treatment Sequence 2: Single subcutaneous (SC) dose of BIIB017 on Day 1; and SC doses of Rebif on Days 29, 32, 34, 36, 39, and 41
  Interventions: Drug: peginterferon beta-1a; Drug: Rebif

INTERVENTIONS:
Drug: peginterferon beta-1a — Administered as subcutaneous injection
  Other Names: BIIB017; Plegridy
Drug: Rebif — Administered as subcutaneous injection

SUMMARY:
The primary outcome of the study is to evaluate the cumulative area under the concentration time curve (AUC) over 2 weeks, as measured by AUC from time 0 to 336 hours post dose (AUC0-336h), for serum concentrations of BIIB017 and Rebif.

The secondary outcomes are to evaluate the maximum observed serum concentrations (Cmax) of BIIB017 and Rebif and to evaluate the safety and tolerability of BIIB017 and Rebif over 2 weeks in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

- Must have a body mass index of 19 to 30 kg/m2, inclusive, and minimum body weight of 45.0 kg at Screening and Day -1

Key Exclusion Criteria:

* History or positive test result at Screening for human immunodeficiency virus, hepatitis C virus antibody or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb])
* History of premalignant and malignant disease including solid tumors and hematologic malignancies
* Known allergy to any interferon or any component of BIIB017
* Prior treatment with any investigational drug within the 30 days prior to Day 1, or within 5 half-lives of the drug, whichever is longer

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cumulative area under the concentration-time curve (AUC), as measured by area under the concentration-time curve from time zero to 336 hours post dose (AUC0-336h) | 2 weeks

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of BIIB017 and Rebif | 2 weeks
Number of participants experiencing Adverse Events (AE) and Serious Adverse Events (SAE) | Up to 4 weeks following treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Evansville, Indiana, United States

REFERENCES:
- [Derived] Hu X, Shang S, Nestorov I, Hasan J, Seddighzadeh A, Dawson K, Sperling B, Werneburg B. COMPARE: Pharmacokinetic profiles of subcutaneous peginterferon beta-1a and subcutaneous interferon beta-1a over 2 weeks in healthy subjects. Br J Clin Pharmacol. 2016 Aug;82(2):380-8. doi: 10.1111/bcp.12968. Epub 2016 May 29. PMID 27060836